CLINICAL TRIAL: NCT00971945
Title: Rollover Study of Weekly Paclitaxel (BMS-181339) in Patients With Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA139-387
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Results first posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; BMS 181339

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paclitaxel (Experimental)
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — Solution, I.V., 100 mg/m2, Weekly for 6 of 7 weeks, Until disease progression or unacceptable toxicity became apparent
  Other Names: Taxol; BMS-181339

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of continued administration of paclitaxel given weekly in subjects considered to need to continue treatment after completion of the preceding "Phase II Clinical Study of Weekly Paclitaxel (BMS-181339) with Advanced Breast Cancer (Protocol No. CA139-371)"

ELIGIBILITY:
Inclusion Criteria:

* Subjects who were confirmed to have a response after receiving at least two courses of weekly paclitaxel therapy and considered to need to continue the therapy by the investigator/subinvestigator among the patients with advanced or recurrent breast cancer who had met the selection criteria and participated in the preceding phase II clinical study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2005-06-30 (Actual); Primary Completion 2008-03-31 (Actual); Study Completion 2008-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- Japan (4):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Hiroshima, Hiroshima
  - Local Institution, Kagoshima, Kagoshima-ken
  - Local Institution, Toshima-ku, Tokyo

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Six participants were enrolled and treated.
Groups:
- Treatment Arm: Paclitaxel 100 mg/m2 IV administered on Days 1, 8, 15, 22, 29, 36 and then suspended until Day 49 (1 course comprised of 49 days).
Period: Overall Study
Arm/Group | Treatment Arm
Started | 6
Completed | 0
Not Completed | 6
Not completed — Progressive Disease | 3
Not completed — Change in treatment policy | 1
Not completed — Other reasons | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: Years] | 46.0 [33 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Adverse Events
Description: This outcome describes the number of participants experiencing any type, any grade, any cause adverse events (assessed both subjectively and objectively)
Time Frame: From first dose to end of follow-up period (up to approximately 33 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 6
Participants | 6

2. Primary Outcome: Number of Participants Experiencing Laboratory Tests Abnormalities
Description: This outcome describes the number of participants experiencing laboratory test abnormalities. The following laboratory test categories were analyzed:
  * Enzyme investigations
  * Hematology investigations
  * Hepatobiliary investigations
  * Lipid investigations
  * Protein and chemistry analyses
  * Renal and urinary tract investigations
  * Water, electrolytes and mineral investigation. Laboratory test abnormalities were graded according to the NCI Common Toxicity Criteria version 2 (JCOG Version), resulting in a score from Grade 0 (Normal) to Grade 5 (Death due to toxicity).
  Only laboratory test abnormalities with a Grade 3 or higher are reported
Time Frame: From first dose to end of follow-up period (up to approximately 33 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 6
Participants
  Hematology investigations | 1
  Lipid analyses | 1

3. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the number (percentage) of participants achieving either a Complete Response (CR) or Partial Response (PR) to therapy. CR is defined as disappearance of all target lesions, while PR is defined as at least a 30% decrease in the sum of longest diameter (LD) of all target lesions (taking as reference the baseline sum LD).
  Target Lesions were evaluated according to "Evaluation Criteria on the Therapeutic Effects in Patients with Advanced or Recurrent Breast Cancer."
Time Frame: From first dose to end of follow-up period (up to approximately 33 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 6
Participants | 5

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the median time from the first date of Partial Response (assessed as per the "Evaluation Criteria on the Therapeutic Effects in Patients with Advanced or Recurrent Breast Cancer") to the first date of Progressive Disease. Participants were evaluated for DOR in 2 separate studies (NCT01023204 and NCT00971945). Results are representative of the cumulative DOR assessed in both studies.
Time Frame: From first date of Partial Response (in study NCT01023204) to first date of Progressive Disease (in study NCT01023204 or NCT00971945) (up to approximately 37 months)
Population: All treated participants (enrolled in study NCT01023204 and NCT00971945) with PR
Measure: Median (Full Range); unit: Days
Arm/Group | Treatment Arm
Number analyzed (Participants) | 6
Days | 840 [229 to 1156]

ADVERSE EVENTS:
Time Frame: From first dose to 14 days following last dose
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=6)
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=6)
Ear pain (Ear and labyrinth disorders) | 1
Adrenal haemorrage (Endocrine disorders) | 1
Lacrimation increased (Eye disorders) | 2
Conjunctival haemorrage (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Xerophthalmia (Eye disorders) | 1
Dacryostenosis acquired (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Oedema (General disorders) | 5
Fatigue (General disorders) | 4
Asthenia (General disorders) | 2
Chest discomfort (General disorders) | 1
Pain (General disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Nasopharyngitis (Infections and infestations) | 4
Cellulitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumonia mycoplasmal (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Purulence (Infections and infestations) | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Wound complication (Injury, poisoning and procedural complications) | 1
Weight increased (Investigations) | 3
Weight decreased (Investigations) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Hypoaesthesia (Nervous system disorders) | 6
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Calculus ureteric (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Residual urine (Renal and urinary disorders) | 1
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1
Breast inflammation (Reproductive system and breast disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 6
Nail disorder (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2005-05-25): https://cdn.clinicaltrials.gov/large-docs/45/NCT00971945/Prot_000.pdf
  • Statistical Analysis Plan (2007-10-16): https://cdn.clinicaltrials.gov/large-docs/45/NCT00971945/SAP_001.pdf